CLINICAL TRIAL: NCT02063113
Title: Vulnerability and Therapeutic Changes in Older Patients With Multiple Myeloma.
Acronym: MYELOME-PA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inclusion difficulty
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC13_0437
Record Dates: First submitted 2014-02-11; First posted 2014-02-14 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Multiple Myeloma in Older Patients
Keywords: Multiple myeloma,; Older patient,; Treatment,; Geriatric assessment
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NA/NA (No Intervention)
  Interventions: Other: Vulnerability and therapeutic changes in older patients with multiple myeloma.

INTERVENTIONS:
Other: Vulnerability and therapeutic changes in older patients with multiple myeloma.

SUMMARY:
The aim of this study is to determine whether the presence of vulnerability detected by geriatricians is associated with treatment discontinuation in older patient. During the comprehensive geriatric assessment realized before the decision-treatment, the following data are recorded and their impact in the therapeutic changes will also be analysed: comorbidity, age, depression, functional status, the cognitive impairment and malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 70 years and older
* Patients referred for a assessment of a newly diagnosed multiple myeloma
* Patients for who the initial therapy proposed is either melphalan-prednisone-thalidomide or melphalan-prednisone-bortezomib or included in a phase 3 trial.
* Patients who provide informed written consent

Exclusion Criteria:

* Patients who refuse the study
* Patients who won't have therapy
* Patients can't respond to geriatric assessment because of severe cognitive disorder
* Patients with a legal guardian

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-05-19 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
The occurrence of the events | 6 MONTHS
  The primary outcome is either :
  * early interruption of treatment
  * dose reduction > 20% during treatment
  * discontinuous treatment
  These outcomes will be measured every 6 months during the 2 years of follow up

SECONDARY OUTCOMES:
Type of Vulnerability | 6 MONTHS
  vulnerability related to toxicities, vulnerability related to multiple myeloma or geriatric vulnerability.
Therapeutic changes | 6 MONTHS
  early interruption of treatment, dose reduction during treatment, discontinuous treatment
Toxicity during treatment | 6 months
  hematologic toxicity, neurotoxicity, gastrointestinal toxicity, deep vein thrombosis, pulmonary embolism, infections with antibiotic use
Progression to 1 and 2 years | 1 year/2year
Complete response at 1 and 2 years | 1 year/2 years

CONTACTS AND LOCATIONS:
Overall Officials: Komivi AGBETSIVI, DR, Principal Investigator — CHD Vendée La Roche sur Yon; VIGNARD Patricia, Dr, Principal Investigator — CH du Mans; Catherine Cattenoz, Dr, Principal Investigator — Rennes University Hospital; Jean -Richard EVEILLARD, Dr, Principal Investigator — CHU de Brest; François Puisieux, Pr, Principal Investigator — CHU de Lille; Jean -Yves NIEMIER, Dr, Principal Investigator — Central Hospital, Nancy, France; Frédérique Retornaz, Dr, Principal Investigator — CGD de Marseille; Véronique Brunel, Dr, Principal Investigator — Hôpital Européen de Marseille; Laure De Decker, Dr, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - CHD Vendée La Roche sur Yon, La Roche-sur-Yon
  - CHU de Nantes, Nantes